CLINICAL TRIAL: NCT04035473
Title: A Randomized Crossover Study to Determine the Bioequivalence of Three Consecutive Daily Doses of Oraxol in Cancer Patients Treated With Intravenous Paclitaxel
Brief Title: A Study to Determine the Bioequivalence of Oraxol in Cancer Patients Treated With Intravenous Paclitaxel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Athenex, Inc. (Industry)
Collaborators: PharmaEssentia (Industry); Zenith Technology Corporation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KX-ORAX-002
Record Dates: First submitted 2019-06-14; First posted 2019-07-29 (Actual); Results first posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-02

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Oraxol, IV paclitaxel) (Active Comparator): The treatment sequences will be:
  A Oraxol (paclitaxel + HM30181) on Days 1, 2, and 3 of Treatment Period 1 followed by IV paclitaxel on Day 1 of Treatment Period 2 B IV paclitaxel on Day 1 of Treatment Period 1 followed by Oraxol on Days 1, 2, and 3 of Treatment Period 2
  Interventions: Drug: HM30181 methanesulfonate monohydrate plus oral paclitaxel capsules
- Sequence B (IV paclitaxel, Oraxol) (Active Comparator): The treatment sequences will be:
  A IV paclitaxel on Day 1 of Treatment Period 1 followed by Oraxol on Days 1, 2, and 3 of Treatment Period 2 B Oraxol (paclitaxel + HM30181) on Days 1, 2, and 3 of Treatment Period 1 followed by IV paclitaxel on Day 1 of Treatment Period 2
  Interventions: Drug: HM30181 methanesulfonate monohydrate plus oral paclitaxel capsules

INTERVENTIONS:
Drug: HM30181 methanesulfonate monohydrate plus oral paclitaxel capsules — HM30181 methanesulfonate monohydrate plus oral paclitaxel capsules
  Oral paclitaxel capsules
  Other Names: ORAXOL

SUMMARY:
This is a multicenter, open-label, 2-stage study with a 2-treatment period crossover design. Eligible participants are adults with cancer for whom weekly therapy with IV paclitaxel at a dose of 80 mg/m2 over 1 hour is indicated.

Stage 1 will consist of an initial cohort (Cohort 1) up to 6 evaluable participants who will receive a dosing regimen of Oraxol consisting of a 15-mg oral HM30181AK-US tablet plus an oral paclitaxel dose of 205 mg/m2, both administered once daily for 3 consecutive days. The stages and cohorts are further described in the "Study Design - Stages and Cohorts" table below. An interim analysis of pharmacokinetic (PK) data from Cohort 1 will be conducted to determine if the administered regimen would appear likely to achieve bioequivalence(BE) (AUC0-∞), if tested in a greater number of participants in Stage 2. If it appears unlikely that the selected regimen will meet the criteria for BE based on AUC0-∞ data, a second cohort (Cohort 2) of up to 6 evaluable participants may be enrolled in Stage 1, and the dose of paclitaxel in Oraxol may be adjusted by a maximum of +/- 25%. If Cohort 2 is enrolled, a second interim analysis will be conducted.

After the interim analysis/analyses (depending on the outcomes), a decision will be made by consensus of the Data Safety and Monitoring Board(DSMB), Kinex, Zenith Technology, and the Principal Investigator as to what dose should be administered in Stage 2. The DSMB will consist of a clinical oncologist, an ethicist, an independent statistician, and additional members, as deemed necessary. A DSMB charter will describe the planned evaluations and decision points used to determine the dose for Stage 2. An additional 18 to 42 evaluable participants will be enrolled into Stage 2 based on the Stage 1 results (AUC0-∞). Thus a total of up to 54 evaluable participants could potentially be enrolled in this study (6 each from Stage 1, Cohorts 1 and 2, and up to 42 participants in Stage 2).

DETAILED DESCRIPTION:
Stage 1 will consist of an initial cohort (Cohort 1) up to 6 evaluable participants who will receive a dosing regimen of Oraxol consisting of a 15-mg oral HM30181AK-US tablet plus an oral paclitaxel dose of 205 mg/m2, both administered once daily for 3 consecutive days. The stages and cohorts are further described in the "Study Design - Stages and Cohorts" table below. An interim analysis of pharmacokinetic (PK) data from Cohort 1 will be conducted to determine if the administered regimen would appear likely to achieve bioequivalence (BE) (AUC0-∞), if tested in a greater number of participants in Stage 2. If it appears unlikely that the selected regimen will meet the criteria for BE based on AUC0-∞ data, a second cohort (Cohort 2) of up to 6 evaluable participants may be enrolled in Stage 1, and the dose of paclitaxel in Oraxol may be adjusted by a maximum of +/- 25%. If Cohort 2 is enrolled, a second interim analysis will be conducted.

After the interim analysis/analyses (depending on the outcomes), a decision will be made by consensus of the Data Safety and Monitoring Board(DSMB), Kinex, Zenith Technology, and the Principal Investigator as to what dose should be administered in Stage 2. The DSMB will consist of a clinical oncologist, an ethicist, an independent statistician, and additional members, as deemed necessary. A DSMB charter will describe the planned evaluations and decision points used to determine the dose for Stage 2. An additional 18 to 42 evaluable participants will be enrolled into Stage 2 based on the Stage 1 results (AUC0-∞). Thus a total of up to 54 evaluable participants could potentially be enrolled in this study (6 each from Stage 1, Cohorts 1 and 2, and up to 42 participants in Stage 2).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Males and females ≥18 years of age on day of consent
3. Cancer patients for whom treatment with IV paclitaxel at 80 mg/m2has been recommended by their oncologist, either as monotherapy or in combination with other agents
4. Adequate hematologic status at Screening/Baseline:

   * Absolute neutrophil count (ANC) ≥1.5 x 109/L
   * Platelet count ≥100 x 109/L
   * Hemoglobin (Hgb) ≥90 g/L
5. Adequate liver function at Screening/Baseline as demonstrated by:

   * Total bilirubin of ≤20 μmol/L or ≤30 μmol/L for participants with liver metastasis
   * Alanine aminotransferase (ALT) ≤3 x upper limit of normal (ULN) or ≤5 x ULN if liver metastasis is present
   * Alkaline phosphatase (ALP) ≤3 x ULN or ≤5 x ULN if liver or bone metastasis are present
   * ALP >5 x ULN if liver or bone metastasis are present and the major fraction of ALP is from bone metastasis, at the discretion of the Investigator
   * Gamma glutamyl transferase (GGT) <10 x ULN
6. Adequate renal function at Screening/Baseline as demonstrated by serum creatinine ≤177 μmol/L or creatinine clearance >50 mL/min as calculated by the Cockcroft and Gault formula
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 16
8. Life expectancy of at least 3 months
9. Willing to fast for 8 hours before and 4 hours after Oraxol administration
10. Willing to abstain from alcohol consumption for 3 days before the first dose of study drug through the completion of protocol-specified PK sampling in Treatment Period 2
11. Willing to refrain from caffeine consumption for 12 hours before each treatment period through the completion of protocol-specified PK sampling for that dose
12. Women must be postmenopausal (>12 months without menses) or surgically sterile (ie, by hysterectomy and/or bilateral oophorectomy) or, if sexually active, must be using effective contraception (ie, oral contraceptives, intrauterine device, double barrier method of condom and spermicide) and agree to continue use of contraception for the duration of their participation in the study. Women of childbearing potential must agree to use contraception for 30 days after their last dose of study drug.
13. Sexually active male participants must use a barrier method of contraception during the study and agree to continue the use of male contraception for at least 30 days after the last dose of study drug.

Exclusion Criteria:

1. Currently taking a prohibited concomitant medication:

   * Strong inhibitors (eg, ketoconazole) or strong inducers (eg, rifampin or St. John's Wort) of cytochrome P450 (CYP) 3A4 (within 2 weeks prior to the start of dosing in the study)
   * Strong inhibitors (eg, gemfibrozil) or strong inducers (eg, rifampin) of CYP2C8 (within 2 weeks prior to the start of dosing in the study)
   * Known P-glycoprotein (P-gp) inhibitors or inducers. Participants who are taking such medications but who are otherwise eligible may be enrolled if they discontinue the medication ≥1 week before dosing and remain off that medication through the end of PK sampling after the administration of the second study treatment.
   * An oral medication with a narrow therapeutic index known to be a P-gp substrate (eg, digoxin, dabigatran) within 24 hours prior to start of dosing in the study
2. Use of warfarin. Participants receiving warfarin who are otherwise eligible and who may be appropriately managed with low molecular weight heparin, in the opinion of the Investigator, may be enrolled in the study provided they are switched to low molecular weight heparin at least 7 days prior to receiving study treatment.
3. Unresolved toxicity from prior chemotherapy (participants must have recovered all significant toxicity to ≤ Grade 1 CTCAE toxicity1 from previous anticancer treatments or previous investigational agents). This does not extend to symptoms or findings that are attributable to the underlying disease
4. Received investigational agents within 14 days or 5 half-lives prior to the first study dosing day, whichever is longer
5. Women of childbearing potential who are pregnant or breastfeeding
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, clinically significant myocardial infarction within the last 6 months, unstable angina pectoris, clinically significant cardiac arrhythmia, bleeding disorder, chronic pulmonary disease requiring oxygen, or psychiatric illness/social situations that would limit compliance with study requirements
7. Major surgery to the upper GI tract, or have a history of GI disease or other medical condition that, in the opinion of the Investigator may interfere with oral drug absorption
8. A known history of allergy to paclitaxel. Participants whose allergy was due to the IV solvent (such as Cremophor®) and not paclitaxel will be eligible for this study.
9. Any other condition which the Investigator believes would make a subject's participation in the study not acceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Cutler, MD, Study Director — Athenex, Inc.
Locations (7):
- Monash Medical Centre, Melbourne, Australia
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Dunedin Hospital, Dunedin
  - Wellington Regional Hospital, Wellington
- Taiwan (3):
  - Shuang Ho hospital, New Taipei City
  - Tri-Service General Hospital, Taipei
  - Lotung Poh-Ai Hospital, Yilan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 45 subjects signed ICF. 3 subjects were screening failures and 42 were randomized. All of the screen failure subjects failed to meet inclusion or exclusion criteria
Groups:
- Sequence A (Oraxol, IV Paclitaxel): Oraxol (15 mg HM30181AK-US tablet + 205 mg/m2 paclitaxel capsules) on Days 1, 2, and 3 of Treatment Period 1 followed by 80 mg/m2 IV paclitaxel on Day 1 of Treatment Period 2
- Sequence B (IV Paclitaxel, Oraxol): 80 mg/m2 IV paclitaxel on Day 1 of Treatment Period 1 followed by Oraxol (15 mg HM30181AK-US tablet + 205 mg/m2 paclitaxel capsules) on Days 1, 2, and 3 of Treatment Period 2
Period: Screening/Baseline
Arm/Group | Sequence A (Oraxol, IV Paclitaxel) | Sequence B (IV Paclitaxel, Oraxol)
Started | 20 | 22
Completed | 20 | 20
Not Completed | 0 | 2
Not completed — Death | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Treatment Period 1
Arm/Group | Sequence A (Oraxol, IV Paclitaxel) | Sequence B (IV Paclitaxel, Oraxol)
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | Sequence A (Oraxol, IV Paclitaxel) | Sequence B (IV Paclitaxel, Oraxol)
Started | 18 (2 subjects withdrew before starting treatment period 2 due to diease progression and withdrawal from study treatment and procedure.) | 19 (1 subject withdrew before starting treatment period 2 due to SAE and investigator's decision.)
Completed | 18 | 19
Not Completed | 0 | 0
Period: Follow-up Period
Arm/Group | Sequence A (Oraxol, IV Paclitaxel) | Sequence B (IV Paclitaxel, Oraxol)
Started | 18 | 19
Completed | 16 | 19
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: Of the 42 randomized subjects, 2 discontinued study participation due to an AE prior to receiving study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A (Oraxol, IV Paclitaxel) | Sequence B (IV Paclitaxel, Oraxol) | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (10.12) | 59.85 (12.14) | 60.33 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 15 | 15 | 30
  Taiwan | 3 | 5 | 8
  Australia | 2 | 0 | 2
Weight [Mean (Standard Deviation); unit: kg] | 70.89 (15.45) | 75.42 (15.32) | 73.16 (15.36)
Height [Mean (Standard Deviation); unit: cm] | 166.13 (8.50) | 166.05 (7.82) | 166.09 (8.06)
Body Surface Area [Mean (Standard Deviation); unit: m^2] | 1.78 (0.20) | 1.84 (0.20) | 1.81 (0.20)
ECOG [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status is a simple measure of functional status. It has scores ranging from 0 to 5. It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability like walking or working. A higher score means a worse functional status. Score 0: Asymptomatic, 1: Symptomatic but completely ambulatory; 2: Symptomatic, <50% in bed during the day; 3: Symptomatic, >50% in bed, but not bedbound; 4: Bedbound; 5: Death.
  Participants
    0 | 8 | 12 | 20
    1 | 12 | 8 | 20
    2 | 0 | 0 | 0
    3 | 0 | 0 | 0
    4 | 0 | 0 | 0
    5 | 0 | 0 | 0
Tumor Stage at Screening [Count of Participants; unit: Participants] — Tumor stage was assessed using the Tumor, Node, Metastasis (TNM) system. Under the TNM staging system, Stage I-III reflect that cancer is present, with the higher the number, the larger the cancer tumor and the more it has spread into nearby tissues. Stage IV indicates that the cancer has spread to distant parts of the body.
  Participants
    Stage II | 1 | 1 | 2
    Stage III | 2 | 0 | 2
    Stage IV | 15 | 17 | 32
    Not Applicable | 2 | 2 | 4
Metastatic Site [Count of Participants; unit: Participants]
  Bone | 9 | 9 | 18
  Kidney | 1 | 0 | 1
  Lungs | 6 | 9 | 15
  Lymph Nodes | 10 | 10 | 20
  Liver | 7 | 8 | 15
  Other | 9 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve Zero Time Extrapolated to Infinite Time (AUC0-∞)
Description: Paclitaxel plasma concentrations were normalized to 615 mg/m2 for Oraxol and 80 mg/m2 for IV paclitaxel.
  Pharmacokinetic and statistical analyses were based on normalized plasma concentrations. Plasma concentrations for paclitaxel were analyzed to determine AUC0-∞ by noncompartmental analysis using plasma concentration-time data for oral and IV paclitaxel
Time Frame: Pharmacokinetic Sampling for IV Paclitaxel - Predose to 96 hours after infusion (Day 1-5). Pharmacokinetic Sampling for Oraxol- predose of Day1 to 144 hours after third dose of day 3 (Day 1-9)
Population: The 35 randomized subjects completed the study and made up the PK Analysis Set
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Oraxol: 615 mg/m2 over 3 Consecutive Days Administered as Oraxol
- IV Paclitaxel: IV paclitaxel (80 mg/m2) infused over 1 hour
Arm/Group | Oraxol | IV Paclitaxel
Number analyzed (Participants) | 35 | 35
ng*h/mL | 5033.5 (1401.1) | 5595.9 (264.1)

2. Secondary Outcome: Maximum Observed Concentration (Cmax)
Description: Paclitaxel plasma concentrations were normalized to 615 mg/m2 for Oraxol and 80 mg/m2 for IV paclitaxel.
  Pharmacokinetic and statistical analyses were based on normalized plasma concentrations. Plasma concentrations for paclitaxel were analyzed to determine Cmax by noncompartmental analysis using plasma concentration-time data for oral and IV paclitaxel
Time Frame: as for outcome 1
Population: The 35 randomized subjects completed the study and made up the PK Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oraxol | IV Paclitaxel
Number analyzed (Participants) | 35 | 35
ng/mL | 397.2 (157.3) | 2732.8 (629.7)

3. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to Time of Last Quantifiable Concentration (AUC0-t)
Description: Paclitaxel plasma concentrations were normalized to 615 mg/m2 for Oraxol and 80 mg/m2 for IV paclitaxel.
  Pharmacokinetic and statistical analyses were based on normalized plasma concentrations. Plasma concentrations for paclitaxel were analyzed to determine AUC0-t by noncompartmental analysis using plasma concentration-time data for oral and IV paclitaxel
Time Frame: as for outcome 1
Population: The 35 randomized subjects completed the study and made up the PK Analysis Set
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Oraxol | IV Paclitaxel
Number analyzed (Participants) | 35 | 35
ng*h/mL | 4829.4 (1375.1) | 5431.8 (1200.3)

4. Secondary Outcome: Time at Which the Highest Drug Concentration Occurs (Tmax)
Description: Paclitaxel plasma concentrations were normalized to 615 mg/m2 for Oraxol and 80 mg/m2 for IV paclitaxel.
  Pharmacokinetic and statistical analyses were based on normalized plasma concentrations. Plasma concentrations for paclitaxel were analyzed to determine Tmax by noncompartmental analysis using plasma concentration-time data for oral and IV paclitaxel
Time Frame: as for outcome 1
Population: The 35 randomized subjects completed the study and made up the PK Analysis Set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Oraxol | IV Paclitaxel
Number analyzed (Participants) | 35 | 35
hours | 1.4 (0.6) | 1.0 (0.2)

5. Secondary Outcome: Terminal Elimination Phase Half-life (t½)
Description: Paclitaxel plasma concentrations were normalized to 615 mg/m2 for Oraxol and 80 mg/m2 for IV paclitaxel.
  Pharmacokinetic and statistical analyses were based on normalized plasma concentrations. Plasma concentrations for paclitaxel were analyzed to determine t½ by noncompartmental analysis using plasma concentration-time data for oral and IV paclitaxel
Time Frame: as for outcome 1
Population: The 35 randomized subjects completed the study and made up the PK Analysis Set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Oraxol | IV Paclitaxel
Number analyzed (Participants) | 35 | 35
hours | 42.8 (8.6) | 26.1 (4.3)

6. Secondary Outcome: Safety and Tolerability of Oraxol Compared With IV Paclitaxel
Description: Safety was assessed by recording all adverse events (AEs) and serious adverse events (SAEs), including CTCAE grades (version 4.03); recording concomitant medications; clinical laboratory testing (including hematology, biochemistry, and urinalysis); measurement of vital signs (pulse rate, systolic and diastolic blood pressures, respiratory rate, and body temperature), weight, and body surface area (BSA); performance of electrocardiograms (ECGs); assessment of ECOG performance status; and performance of physical examinations
Time Frame: From screening until final visit (within 28 days after the last dose of study drug was taken, and preferably before the participant receives any additional chemotherapy)
Population: 40 subjects received study drug (39 received at least 1 dose of Oraxol and 38 received 1 dose of IV paclitaxel) and had at least 1 postdose safety assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Oraxol | IV Paclitaxel
Number analyzed (Participants) | 39 | 38
Participants
  TEAE | 36 | 29
  Treatment-related TEAE | 30 | 20
  Grade 3 TEAE | 7 | 2
  TEAE leading to study drug discontinuation | 1 | 2
  TEAE leading to study discontinuation | 0 | 2
  TEAE resulting in death | 0 | 1

ADVERSE EVENTS:
Time Frame: up to 7 weeks
Groups:
- Oraxol: Oraxol (15 mg HM30181A + oral paclitaxel 205 mg/m2) for 3 consecutive days.
- IV Paclitaxel: IV Pacllitaxel 80 mg/m2 for 1 day.
Arm/Group | Oraxol | IV Paclitaxel
All-Cause Mortality (participants affected / at risk) | 0/39 | 1/38
Serious Adverse Events (participants affected / at risk) | 4/39 | 2/38
Other Adverse Events (participants affected / at risk) | 36/39 | 29/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oraxol (N=39) | IV Paclitaxel (N=38)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oraxol (N=39) | IV Paclitaxel (N=38)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 7 (7)
Nausea (Gastrointestinal disorders) | 11 (11) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (6) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (6) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 1 (2)
Injection site pruritus (General disorders) | 1 (1) | 0 (0)
Medical device site irritation (General disorders) | 0 (0) | 1 (1)
Medical device site rash (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 2 (3) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dysphonia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 5 (5)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood calcium increased (Investigations) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT04035473/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT04035473/SAP_001.pdf